CLINICAL TRIAL: NCT06111105
Title: GUIding Multi-moDal ThErapies Against MRD by Liquid Biopsies in Colorectal Cancer - GUIDE.MRD-01-CRC
Brief Title: GUIDE.MRD-01-CRC: Clinical Validation and Benchmarking of Top Performing CtDNA Diagnostics - Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Claus Lindbjerg Andersen (Other)
Collaborators: Medical University of Graz (Other); University Medical Centre of Montpellier (Unknown); Universitätsklinikum Hamburg-Eppendorf (Other); University of Aarhus (Other); Karolinska Institutet (Other)
Responsible Party: Sponsor-Investigator, Claus Lindbjerg Andersen, Professor, University of Aarhus
Organization: University of Aarhus (Other)
Other Study IDs: GUIDE.MRD-01-CRC
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer Stage III; Liver Metastasis Colon Cancer
Keywords: Circulating tumor DNA; ctDNA diagnostics; Minimal residual disease
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Full blood samples processed into plasma, buffy coat, and serum Formalin-fixed paraffin-embedded tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Colorectal cancer stage III
- Colorectal cancer liver metastasis

SUMMARY:
Improving personalized cancer treatments and finding the best strategies to treat each patient relies on using new diagnostic technologies. Currently, for colorectal cancer, the methods used to decide who gets additional post-surgery treatment are suboptimal. Some patients get too much treatment, while others do not get enough.

There is a new way to explore if there is any cancer left in a patient's body using circulating tumor DNA (ctDNA) detected in blood samples. This can help decide who needs more treatment after surgery. Even though many tests have been developed, it has yet to be determined which test performs best at relevant time points.

The GUIDE.MRD consortium is a group of experts, including scientists, technology, and pharmaceutical companies. The consortium is working on creating a reliable standard for the ctDNA tests, validating their clinical utility, and collecting data to help decide on the best treatment for each patient.

GUIDE.MRD-01-CRC is a part of the GUIDE.MRD project.

DETAILED DESCRIPTION:
GUIDE.MRD-01-CRC is a part of WP3 of the overarching GUIDE.MRD project. Each study chair has a local clinical trial protocol where patients are recruited. After the end of recruitment, samples will be analyzed under the GUIDE.MRD consortium.

The overall aim of GUIDE.MRD is to investigate the clinical utility of ctDNA analysis to predict and guide the choice of multi-modal therapies prospectively. The fundamental steps towards this aim are assessment and benchmarking of the many available ctDNA diagnostics to identify the best-suited tests for clinical application. Clinical samples will be used to benchmark ctDNA diagnostics and assess their true clinical performance. The samples should reflect clinical situations where the ctDNA diagnostics are particularly useful, such as post-operatively, post-adjuvant, during chemotherapy, and longitudinally during post-treatment surveillance. In these situations, ctDNA diagnostics could be used to either monitor treatment response (in case of MRD after surgery) or to identify relapse at an early time point. Based on ctDNA information, medical treatment could be changed, or radiology could be used to reveal the location of residual disease.

The rationale for the observational clinical study GUIDE.MRD-01-CRC is to prospectively collect the clinical samples needed to enable assessment of the performance of ctDNA diagnostics in the setting of colorectal cancer (CRC). There are two main scenarios where ctDNA diagnostic is useful in CRC:

Stage III CRC (locally advanced, non-metastasized disease): This patient group is particularly relevant because adjuvant therapy is recommended for all stage III patients, due to their high recurrence risk, ~25%. Nevertheless, most patients do not recur, and most of these do not need therapy at all, because they were already cured by surgery alone, which leads to substantial overtreatment. Furthermore, the 25% of patients who recur despite both surgery and adjuvant therapy, probably could benefit from further multimodal therapies. The challenge is, however, that currently there is no marker in clinical use that can identify those patients with residual disease and need for therapy. Circulating tumor DNA is potentially such a marker. However, currently, it is unknown, which, if any, of the many different ctDNA diagnostics developed in recent years have the required performance to provide clinical utility in the management of stage III CRC. This clinical dilemma will be addressed with the first cohort of GUIDE.MRD-01-CRC.

Metastatic CRC with isolated liver metastases. Metastatic CRC with liver metastases is a unique tumor type in that surgical resection or complete ablation of the metastases, is the standard of care. In virtually all other tumor types, resection of liver metastases is considered only within clinical trials or in exceptional clinical circumstances. In contrast, resection, or ablation of colorectal cancer liver metastases (CRLM) are routinely performed with curative intention, and the overall 5-year survival is around 50%. Most relapses present within three years after operative intervention. The clinical benefit of adjuvant chemotherapy is currently a matter of debate, due to limited data from randomized controlled trials and recent results that indicate inferior overall survival (OS) in patients who received adjuvant therapy (JCOG0603). Based on these and earlier data (EORTC Trial 40983) that failed to show an OS benefit of adjuvant therapy after CRLM resection, it can be assumed that most patients are treated unnecessarily with chemotherapy, and those patients that could receive targeted agents are missed. No histological or clinical markers are available to guide decisions on adjuvant treatment. In this setting, ctDNA could be valuable to guide decisions on adjuvant chemotherapy (yes/no), the addition of biologicals such as anti-VEGF and anti-EGFR agents, targeted therapies in the case of BRAF mutations, or the presence of microsatellite instability (MSI), for example.

Primary objectives:

* To assess the performance of ctDNA diagnostics using samples collected at the two-landmark time-points "post-surgery" and "post-adjuvant therapy". Sensitivity, specificity, and positive and negative predictive values of the ctDNA diagnostics will be determined to enable a head-to-head performance assessment and benchmarking of ctDNA diagnostics

Secondary objectives

* To assess the ctDNA stratified 3-year recurrence-free survival (RFS)
* To assess the lead time between ctDNA detection and clinical recurrence
* To assess the capacity of the ctDNA diagnostics to predict response to adjuvant therapy

ELIGIBILITY:
Colorectal cancer stage III

Inclusion Criteria:

* Colorectal cancer, UICC stage III
* Has received curative-intent resection and is a candidate for adjuvant chemotherapy
* Patient able to understand and sign written informed consent

Exclusion Criteria:

* Hereditary colorectal cancer linked to familial colonic polyposis or Lynch syndrome
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Verified distant metastases
* Not treated with adjuvant chemotherapy despite indication (incomplete treatment not included)
* Treated with neoadjuvant chemo-radiation therapy
* No tissue sample available for the project, or tumor content in the tissue sample is <20%
* Synchronous colorectal and non-colorectal cancer diagnosed per operative (except skin cancer other than melanoma)
* Other cancers (excluding colorectal cancer or skin cancer other than melanoma) within 3 years from eligibility screening
* Patients who are unlikely to comply with the protocol (e.g. uncooperative attitude), inability to return for subsequent visits) and/or otherwise considered by the Investigator to be unlikely to complete the study

Colorectal cancer liver metastasis

Inclusion Criteria:

* Colorectal cancer liver metastasis
* Planned for curative-intent treatment
* Performance status 0-1

Exclusion Criteria:

* Liver cirrhosis
* Extrahepatic metastases
* Other cancer within the last 5 years
* Intervention not performed with curative intent
* No tissue available from CRLM or primary tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal cancer stage III: patient with stage III colorectal cancer treated with curative-intent surgery and adjuvant chemotherapy
  Colorectal cancer liver metastasis: patient with colorectal cancer liver metastasis
Sampling Method: Non-Probability Sample
Enrollment: 590 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Collection of clinical plasma samples at relevant time points | 8 months after end of recruitment
  For head-to-head performance assessment and benchmarking of ctDNA diagnostics

SECONDARY OUTCOMES:
The 3-year recurrence-free survival | 3 years after end of recruitment
Lead time between ctDNA detection and clinical recurrence | 3 years after end of recruitment
Prognostic value of ctDNA analysis at relevant time points | 3 years after end of recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Heitzer, PhD, Study Chair — Medical University of Graz; Klaus Pantel, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf; Catherine Alix-Panabiéres, PhD, Study Chair — University Medical Centre of Montpellier; Matthias Löhr, MD, Study Chair — Karolinska Institutet; Claus L Andersen, PhD, Study Director — Aarhus University Hospital
Locations (15):
- Austria (2):
  - Abteilung für Onkologie, Medizinische Universität Graz, Graz, Styria
  - Ordenskrankenhaus Graz Mitte, Graz, Styria
- Denmark (9):
  - Bispebjerg Hospital, Copenhagen, Capital Region of Denmark
  - Herlev Hospital, Herlev, Capital Region of Denmark
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Gødstrup Hospital, Herning, Central Jutland
  - Regional Hospital Horsens, Horsens, Central Jutland
  - Regional Hospital Randers, Randers, Central Jutland
  - Regional Hospital Viborg, Viborg, Central Jutland
  - Aalborg University Hospital, Aalborg, North Denmark
  - Odense University Hospital, Odense, The Region of Southern Denmark
- LCCRH (Laboratoire Cellules Circulantes Rares Humaines) - CHU de Montpellier, Montpellier, France
- Germany (2):
  - Department of General-, Visceral- and Thoracic Surgery, University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

REFERENCES:
- See also: Webpage of the GUIDE.MRD project — https://www.guidemrd-horizon.eu/